CLINICAL TRIAL: NCT06756685
Title: Effects of Core Strengthening Versus Motor Control Training on Pain, Disability & Endurance in Patients With Low Back Pain
Brief Title: Effects of Core Strengthening Versus Motor Control Training on Pain, Disability & Endurance in Low Back Pain
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Riphah International University (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Treatment
Other Study IDs: 014384/Sabiha Fayyaz
Record Dates: First submitted 2024-08-13; First posted 2025-01-03 (Actual); Last update posted 2025-08-29 (Actual); Status verified 2025-08

CONDITIONS: Low Back Pain
Keywords: back pain; disability; endurance; core strengthening; motor control
MeSH Terms: conditions — Low Back Pain; Back Pain

STUDY DESIGN:
Who Masked: Participant, Outcomes Assessor
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Core Strengthening Exercises (Experimental): Core Strengthening Exercises
  Interventions: Other: Core Strengthening Exercises
- Motor Control Training (Active Comparator): Motor Control Training
  Interventions: Other: Motor Control Training

INTERVENTIONS:
Other: Core Strengthening Exercises — The Core Strengthening Program participants will have supervised gym-based sessions for 8 weeks. In the first 4 weeks , participants will attend two 1 hour training sessions, followed by self-selected one or two sessions per week. The session will begin with 20min of aerobic conditioning of walking or running on a treadmill, starting at 65% and moving to 85% of HR max. The 5 key elements of focus are i. Centering ii. Breathing iii. Head and neck placement iv. Shoulder placement v. Chest wall placement
  Arms: Core Strengthening Exercises
Other: Motor Control Training — Participants in Motor Control group will receive two physiotherapy sessions of 1hour / week in the first 4 weeks, during stage 1. i. Abdominal drawing-in maneuver (ADIM) : isometric contraction of the local stability muscles (e.g., lumbar multifidus, transversus abdominis) in minimally loading positions (supine lying, quadruped, sitting, and standing) by maintaining a neutral spine while maintaining normal breathing. During Phase 2, One 1 hour session / week in the second 4 weeks.
  Activation and facilitation of transversus abdominis, lumbar multifidus and pelvic floor motor control(36).Exercises target the transversus abdominis, multifidus and pelvic floor muscles plus postural correction to restore optimal motor control during non-weight-bearing activities. Exercises and progressions will follow previous protocols of motor control exercise.
  Arms: Motor Control Training

SUMMARY:
The study aims to compare the effects of core strengthening versus motor control training on pain, disability & endurance in patients with low back pain

DETAILED DESCRIPTION:
The study aims to compare the effects of core strengthening versus motor control training on pain, disability & endurance in patients with low back pain.

Comparing core strength and conditioning versus motor control for low back pain on physical and self-report outcomes lies in identifying the most effective treatment approach for this condition. This will help to determine which one yields better results in terms of improving physical function and reducing self-reported pain and disability associated with low back pain. This study can provide valuable insights for clinicians and patients in selecting the most appropriate treatment option.

ELIGIBILITY:
Inclusion Criteria:

* Non-specific Chronic low back pain (>3 months)
* Pain between the T12 vertebra and gluteal fold with pain of 2-8 on the numerical rating scale of 0-10
* Both Genders
* Age of 25 and above

Exclusion Criteria:

* Participants fall in this category would be excluded of the study.

  * Lumbar radiculopathy
  * Structural scoliosis
  * Traumatic spinal injury
  * Cauda equina syndrome
  * History of seizures, epilepsy, stroke or head injury
  * Metal implants
  * Pregnancy or considering pregnancy in near future
  * Body mass >/= 100kg

Ages: 25 Years to 60 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult
Enrollment: 74 (Actual)
Dates: Start 2024-08-07 (Actual); Primary Completion 2025-01-01 (Actual); Study Completion 2025-01-10 (Actual)

PRIMARY OUTCOMES:
Goniometer | 8 weeks
  A goniometer will be used to measure ranges of motion of Trunk in Flexion, Extension, lateral Flexion and Rotation
Lower body strength | 8 weeks
  One-repetition maximum (1-RM) leg press at 70% 1-RM will be used to evaluate lower body strength.
Modified Oswestry disability index | 8 weeks
  The Oswestry Disability Index is considered one of the best accepted tools for assessment of low back pain. It is a patient-completed questionnaire which gives a subjective percentage score of level of function (disability) in activities of daily living in chronic low back pain. The ODI is made up of 10 items. Each item consist of 6 statements which are scored from 0 to 5. With 0 indicating the least disability and 5 the greatest then the total score is calculated as a percentage, with 0% indicating no disability and 100% indicating the highest level of disability.
  ODI = (Sum of items scored/Sum of sections answered) X 100
Tampa scale of kinesiophobia | 8 weeks
  The Tampa Scale of Kinesiophobia (TSK) was first developed in 1991 by R. Miller, S. Kopri, and D. Todd. A self-reported questionnaire that quantifies fear of movement, or (re)injury.It uses a 4-point Likert scale (Strongly Disagree-Disagree-Agree-Strongly Agree).The 17 item TSK total scores range from 17 to 68 where the lowest 17 means no or negligible kinesiophobia, and the higher scores indicate an increasing degree of kinesiophobia.Scores above 37 (17-item) are generally considered to indicate kinesiophobia.
Visual analog scale | 8 weeks
  The pain VAS is a uni dimensional measure of pain intensity, used to record patients' pain progression, or compare pain severity.Using a ruler, the score is determined by measuring the distance (mm) on the 10-cm line between the "no pain" anchor and the patient's mark, providing a range of scores from 0-100. A higher score indicates greater pain intensity.no pain (0-4 mm), mild pain(5-44 mm), moderate pain (45-74 mm), and severe pain (75-100 mm).Test-retest reliability has been shown to be good and moderate to good reliability for disability in patients with chronic musculoskeletal pain.
Japanese orthopedic association back pain evaluation questionnaire | 8 weeks
  The JOABPEQ includes twenty-five questions that are subdivided into five sub scales: lower back pain, lumbar function, walking ability, social life function, and mental health. These questions are Intended to evaluate individuals with low back pain from five different perspectives.scores range from 0 to 100, with higher scores indicating a better patient condition. Both kappa and weighted kappa were more than 0.50 for all but one item, which was 0.48.

CONTACTS AND LOCATIONS:
Overall Officials: Sabiha Fayyaz, MS-NMPT*, Principal Investigator — Riphah International University
Locations (1):
- Mediplex Health Care Center, Rawalpindi, Punjab Province, Pakistan

IPD SHARING:
Plan to Share IPD: No